CLINICAL TRIAL: NCT02758886
Title: Pet Your Stress Away Study
Acronym: PYSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13711
Record Dates: First submitted 2016-04-12; First posted 2016-05-03 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stress reduction method (Experimental): Participants randomized into the PYSA group engaged in a 10 minute direct interaction with the animals (dogs and cats) of the Pet Your Stress Away program
  Interventions: Behavioral: Animal assisted activity
- Control (Placebo Comparator): Participants randomized into the Control group watched a 10 minute slide show of dog and cat photos
  Interventions: Behavioral: Animal photos
- Non-treatment (No Intervention): Participants randomized into the No-treatment group silently waited for 10 minutes without engaging in any physical or electronic social interactions.
- Observation (Placebo Comparator): Participants randomized into the observation group observed 10 minutes of others in the general PYSA program petting cats and dogs, while they 'waited in line' for there turn.
  Interventions: Behavioral: Observing human-animal interaction

INTERVENTIONS:
Behavioral: Animal assisted activity — Allowed to interact (e.g. talking, petting, scratching, feeding treats, playing with) live animals
  Arms: Stress reduction method
Behavioral: Animal photos — A 10 minute, silent, PowerPoint slide show of a variety of dogs and cats
  Arms: Control
Behavioral: Observing human-animal interaction — Participants watched others participate in petting dogs and cats, while they waited in line for 10 minutes. Participants did not physically touch any animals during this time.
  Arms: Observation

SUMMARY:
The purpose of this study is to determine whether an animal visitation programs on college campuses are effective in the treatment of college student stress reduction during preparation for final examinations.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate status

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in physiological stress measured via salivary cortisol | On the day of program participation: Once immediately upon waking up, and immediately before and after participation in the assigned 10 minute intervention
  Salivary cortisol was measured three times on the day of program participation: immediately upon waking, and immediately before and after participation in the assigned 10 minute intervention
Change in momentary emotion using the experience sampling method questionnaire | Momentary emotion was measured twice, immediately before and after participation in the assigned 10 minute intervention

SECONDARY OUTCOMES:
Change in physiological stress measured via salivary Alpha-amylase | On the day of program participation: Once immediately upon waking up, and immediately before and after participation in the assigned 10 minute intervention
  Salivary alpha-amylase was measured three times on the day of program participation: immediately upon waking, and immediately before and after participation in the assigned 10 minute intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pendry, PhD, Principal Investigator — Washington State University

IPD SHARING:
Plan to Share IPD: No